CLINICAL TRIAL: NCT00479817
Title: A Randomized, Double-Blind, Placebo Controlled, Phase 2 Trial of Paclitaxel in Combination With AMG 386 in Subjects With Advanced Recurrent Epithelial Ovarian or Primary Peritoneal Cancer
Brief Title: Phase 2 AMG 386 in Comb. Paclitaxel for Subjects With Advanced Recurrent Epithelial Ovarian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060342
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Advanced Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — trebananib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): Paclitaxel 80 mg/m2 IV QW (3 on/1 off) + AMG 386 10 mg/kg IV QW
  Interventions: Drug: AMG 386; Drug: Paclitaxel
- Arm B (Experimental): Paclitaxel 80 mg/m2 IV QW (3 on/1 off) + AMG 386 3 mg/kg IV QW
  Interventions: Drug: AMG 386; Drug: Paclitaxel
- Arm C (Active Comparator): Paclitaxel 80 mg/m2 IV QW (3 on/1 off) + AMG 386 placebo
  Interventions: Drug: Paclitaxel; Drug: AMG 386 Placebo

INTERVENTIONS:
Drug: AMG 386 — 10mg/kg
  Arms: Arm A
Drug: AMG 386 — 3 mg/kg
  Arms: Arm B
Drug: Paclitaxel — Paclitaxel 80 mg/m2 IV QW (3 on/1 off)
Drug: AMG 386 Placebo — AMG 386 Placebo
  Arms: Arm C

SUMMARY:
This study is a phase 2, randomized, double-blind, placebo controlled, multi-center study to estimate the improvement in PFS (compared to control subjects) and evaluate the safety and tolerability of AMG 386 in combination with paclitaxel in the treatment of subjects with advanced recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer.

Primary Outcome Measure:

• Progression free survival (PFS)

Secondary Outcome Measures:

* Object Response Rate (ORR), duration of response (DOR). CA-125 response rate
* Safety and Tolerability
* Change and duration of change on blood levels of CA-125

DETAILED DESCRIPTION:
Primary Objective:

To estimate the treatment effect as measured by progression free survival (PFS) of subjects with recurrent ovarian cancer receiving AMG 386 (either 3 mg/kg or 10 mg/kg IV QW) in combination with paclitaxel (80 mg/m2 IV QW; 3 on/1 off)compared to subjects receiving paclitaxel (80 mg/m2 IV QW; 3 on/1 off) plus placebo

Secondary Objective(s):

* To evaluate the safety and tolerability of the combination regimen of AMG 386/paclitaxel
* To estimate other measures of treatment effect (by parameters other than PFS) of subjects receiving AMG 386 in combination with paclitaxel compared to subjects receiving paclitaxel plus placebo
* To evaluate the AMG 386 pharmacokinetics parameters (Cmax and Cmin ) when administered with paclitaxel in subjects with recurrent ovarian cancer
* To estimate the incidence of occurrence of anti-AMG 386 antibody formation
* To estimate the change and duration of change on blood levels of CA-125
* To evaluate the clinical benefit among subjects receiving AMG 386 10 mg/kg monotherapy after disease progression on paclitaxel
* To estimate the impact of AMG 386 on patient reported ovarian cancer specific symptoms and HRQoL using the FACT-O, the FACT-O ovarian cancer subscale (OCS), and the FACT-O 3-item (O1, O2, O3) cancer symptom specific subscale (OCS 3-item subscale)

Exploratory Objective(s):

* To explore the associations between progression free survival, objective response, CA-125, and continuous measures of tumor burden (the percentage change from baseline in the sum of the longest diameters of target lesions)
* To explore the pharmacodynamic (PD) response as assessed by changes in blood levels of angiogenic cytokines, tumor apoptosis, CA-125 and other markers
* To investigate the effects of genetic variation in drug metabolism, cancer genes and drug target genes on ovarian cancer and subject response to investigational product (separate informed consent)
* To explore the impact of AMG 386 on patient reported overall health status as measured by the EuroQoL (EQ-5D)

Hypothesis:

This study will provide an estimate and corresponding 2-sided 80% confidence interval with an approximate maximum half-width of 0.22 of the efficacy, as measured by the PFS hazard ratio of AMG 386 in combination with paclitaxel versus paclitaxel alone for 2 pooled dose groups of AMG 386 (10 mg/kg QW and 3 mg/kg QW) in combination with paclitaxel versus the paclitaxel plus placebo group.

ELIGIBILITY:
In. Criteria -Subjects must have histologically or cytologically documented epithelial ovarian (FIGO Stage II-IV), fallopian tube or primary peritoneal cancer.

(Subjects with pseudomyxoma or mesothelioma are excluded)

* Radiographically documented progression per RECIST criteria with modifications or progression of CA-125 as defined by the Rustin during or subsequent to the last chemotherapy regimen.
* May include measurable or non-measurable disease
* All scans and x-rays used to document measurable or non-measurable disease must be done within 3 weeks (21 days) of enrollment.
* No more than 3 previous regimens of anti-cancer therapy. Subjects must have received at least one platinum containing regimen
* Female 18 years of age or older at the time the written informed consent is obtained
* Subjects of child-bearing potential who have not undergone a bilateral salpingo-oophorectomy and are sexually active must use an accepted and effective non-hormonal method of contraception (ie, double barrier method (eg, condom plus diaphragm)) from signing the informed consent through 6 months after last dose of study drug.

Laboratory

* Adequate organ and hematological function as evidenced by the following laboratory studies within 2 weeks (14 days) of randomization:
* Hematological function, as follows:

Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L and ≤ 850 x 109/L Hemoglobin ≥ 9 g/dL PTT or aPTT≤ 1.5 x ULN per institutional laboratory rand and INR ≤ 1.5 x 109/L per instiutiona laboratory range

Renal function, as follows:

Creatinine ≤ 2.0 mg/dL Calculated creatinine clearance > 40 cc/min according to the Cockcroft-Gault formula

-Hepatic function, as follows: Total bilirubin ≤ 2.0 x ULN SGOT (AST) and SGPT (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present) Nutritional

* Albumin ≥ 2.8 mg/dL General
* GOG Performance Status of 0 or 1
* Subject plans to begin protocol directed therapy within 7 days of randomization Ex Criteria
* Subjects believed to be a higher than average risk for bowel perforation. This includes symptoms of partial or complete bowel obstruction, recent (within 6 months) history of fistula or bowel perforation, subjects requiring total parenteral nutrition and continuous hydration
* Known ongoing small bowel dysfunction (ie, persistent nausea, vomiting)
* Radiotherapy ≤ 14 days prior to randomization. Subjects must have recovered from all radiotherapy-related toxicities
* If all sites of disease have been irradiated, documented progression must have occurred in at least one site of disease subsequent to the radiation therapy.
* Previous abdominal radiotherapy
* Has not yet completed a 21 day washout period for any previous anti-cancer systemic therapies (60 days for bevacizumab or any molecule of long half-life).
* Enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or is receiving other investigational agent(s)
* Current or prior history of central nervous system metastasis
* Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 peripheral neuropathy ≥grade 2
* History of arterial or venous thrombosis within 12 months prior to randomization
* Concurrent or prior (within 1 week before study day 1) anticoagulation therapy, excluding aspirin and anti platelet agents. The concurrent use of low molecular weight heparin or low dose warfarin (ie, ≤ 1 mg daily) for prophylaxis against thrombosis is acceptable while on study
* History of bleeding diathesis or clinically significant bleeding within 14 days of randomization
* Major surgical procedure within 4 weeks (28 days) prior to Study Day 1
* Minor surgical procedure, or placement of central venous access device, within 7 days of Study Day 1
* Paracentesis and/or thoracentesis are permitted prior to and while on study at the discretion of the investigator as clinically indicated. Investigators should document the frequency of paracenteses and/or thoracentesis that occurred prior to the enrollment of the subject in this study on the appropriate eCRFs. Investigators should also document each paracentesis and/or thoracentesis that occurs while a subject is on study on the appropriate eCRFs.
* Subjects with a history of prior malignancy, except:
* Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by treating physician
* Adequately treated non melanomatous skin cancer or lentigo maligna without evidence of disease
* Adequately treated cervical carcinoma in situ without evidence of disease
* Prior myeloablative high dose chemotherapy with allogeneic or autologous stem cell (or bone marrow) transplant
* Clinically significant cardiac disease within 12 months of study enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent
* Non-healing wound, ulcer or fracture
* Ongoing or active infection
* Unacceptable hypersensitivity to paclitaxel or drugs containing cremophor
* Known positive test for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B surface antigen
* Currently or previously treated with angiopoietin inhibitors, or inhibitors of TIE-1 or TIE-2 including, but not limited to, AMG 386, XL880, XL820
* Prior therapy against vascular endothelial growth factor or the vascular endothelial growth factor receptors including, but not limited to, bevacizumab, sunitinib, sorafenib, motesanib (AMG 706) or cediranib (AZD-2171), is permitted so long as the agent does not have any known activity against angiopoietin 1 or 2, or the receptors TIE-1 or TIE-2
* Current or within 30 days of randomization treatment with immune modulators such as cyclosporine and tacrolimus

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2009-08-11 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years

SECONDARY OUTCOMES:
Safety and Tolerability | 2 years
Objective Response Rate | 2 years
Duration of Response | 2 years
Modified RECIST/CA-125 Progression Free Survival | 2 years
CA-125 Response Rate | 2 years
Estimate of reduction in tumor burden | 2 years
Incidence of AEs and significant laboratory changes | 2 years
Overall Survival | 2 years
Time to Progression | 2 years
Time to Response | 2 years
Change from baseline in blood levels of CA-125 | 2 years
Time-adjusted area under the curve for PROs | 2 years
AMG 386 Pharmacokinetic parameters | 2 years
Incidence of the occurence of AMG 386 Antibody formation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Karlan BY, Oza AM, Richardson GE, Provencher DM, Hansen VL, Buck M, Chambers SK, Ghatage P, Pippitt CH Jr, Brown JV 3rd, Covens A, Nagarkar RV, Davy M, Leath CA 3rd, Nguyen H, Stepan DE, Weinreich DM, Tassoudji M, Sun YN, Vergote IB. Randomized, double-blind, placebo-controlled phase II study of AMG 386 combined with weekly paclitaxel in patients with recurrent ovarian cancer. J Clin Oncol. 2012 Feb 1;30(4):362-71. doi: 10.1200/JCO.2010.34.3178. Epub 2011 Dec 19. PMID 22184370
- [Background] Lu JF, Rasmussen E, Karlan BY, Vergote IB, Navale L, Kuchimanchi M, Melara R, Stepan DE, Weinreich DM, Sun YN. Exposure-response relationship of AMG 386 in combination with weekly paclitaxel in recurrent ovarian cancer and its implication for dose selection. Cancer Chemother Pharmacol. 2012 May;69(5):1135-44. doi: 10.1007/s00280-011-1787-5. Epub 2012 Jan 1. PMID 22210018
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com